CLINICAL TRIAL: NCT00636181
Title: Positive Airway Pressure Initiation: Impact of Therapy Mode and Titration Process on Adherence and Outcomes
Brief Title: Positive Pressure Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Principal Investigator, Clete Kushida, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTG3
Record Dates: First submitted 2008-02-06; First posted 2008-03-14 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Auto Aflex (Active Comparator): auto adjusting positive pressure therapy with AFLEX
  Interventions: Device: Auto AFlex
- Auto CPAP (Active Comparator): auto adjusting positive pressure therapy
  Interventions: Device: Auto CPAP
- CPAP (Active Comparator): continuous positive airway pressure
  Interventions: Device: CPAP

INTERVENTIONS:
Device: Auto AFlex — Positive pressure therapy treatment
  Arms: Auto Aflex
Device: Auto CPAP — Positive pressure therapy treatment
  Arms: Auto CPAP
Device: CPAP — Positive pressure therapy treatment
  Arms: CPAP

SUMMARY:
Six month at home positive pressure therapy study; which mode of therapy will lead to better adherence and patient outcomes?

DETAILED DESCRIPTION:
Three arm randomized controlled trial evaluating therapy titration methodologies and device comfort.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 75
* Diagnosis of OSAHS with baseline AHI (Apnea-Hypopnea Index) equal or greater than 15 events/hr of sleep
* Able and willing to provide written informed consent
* Agreement to try PAP (positive airway pressure) as initial treatment approach
* Adequate clinical CPAP titration within two weeks of enrollment

Exclusion Criteria:

* Participation in another interventional research study within the last 30 days
* The need for more than one titration PSG (polysomnography)
* The use of sedatives or hypnotics during the titration PSG
* Major medical or psychiatric condition that would interfere with the demands of the study, adherence to PAP or the ability to commit to follow-up assessment.
* Prior prescription for, or exposure to PAP therapy within the previous year (except exposure to CPAP during clinical therapy titration.)
* Chronic respiratory failure or insufficiency with suspected or known neuromuscular disease, moderate or severe COPD (chronic obstructive pulmonary disease) or other pulmonary disorders, or any condition with an elevation of arterial carbon dioxide levels (>45 mmHG) while awake or participants qualifying for oxygen therapy (arterial saturation < or equal to 88% for more than five minutes).
* Surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days
* Surgery at any time for the treatment of OSAHS such as uvulopalatopharyngoplasty (UPPP)
* Presence of untreated or poorly managed, non-OSAHS related sleep disorders:

  * moderate to severe periodic limb movements (greater or equal to 15 per hour with symptoms or arousals)
  * Restless Leg syndrome (greater than 10 per hour)
  * Males experiencing chronic insomnia
* Use of medications with hypnotic or sedative effects or regular use of night time sedatives or sleeping aids greater than or equal to one night per week.
* Consumption of ethanol more than 4 nights per week (CAGE criteria)
* Shift workers

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clete A. Kushida, M.D.; Ph.D;, Principal Investigator — Stanford University
Locations (5):
- United States (4):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Stanford University, Stanford, California
  - Gaylord Hospital, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
- Charite Universitatsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Aloia MS, Stanchina M, Arnedt JT, Malhotra A, Millman RP. Treatment adherence and outcomes in flexible vs standard continuous positive airway pressure therapy. Chest. 2005 Jun;127(6):2085-93. doi: 10.1378/chest.127.6.2085. PMID 15947324
- [Derived] Kushida CA, Berry RB, Blau A, Crabtree T, Fietze I, Kryger MH, Kuna ST, Pegram GV Jr, Penzel T. Positive airway pressure initiation: a randomized controlled trial to assess the impact of therapy mode and titration process on efficacy, adherence, and outcomes. Sleep. 2011 Aug 1;34(8):1083-92. doi: 10.5665/SLEEP.1166. PMID 21804670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who completed routine clinical diagnostic visit and CPAP titration polysomnography (PSG) at 5 international sleep centers were consecutively recruited for the study. These patients were approached with information on the study and were asked to consent to participate.
Pre-assignment Details: 168 participants were enrolled into the study. However 4 participants were excluded from the analysis and demographic data because they withdrew from the trial prior to any study procedures.
Period: Overall Study
Arm/Group | Auto Aflex | Auto CPAP | CPAP
Started | 54 | 53 | 57
Completed | 46 | 47 | 47
Not Completed | 8 | 6 | 10
Not completed — Withdrawal by Subject | 8 | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auto Aflex | Auto CPAP | CPAP | Total
Number analyzed (Participants) | 54 | 53 | 57 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.6) | 48.3 (10.0) | 48.8 (12.0) | 48.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 14 | 40
  Male | 41 | 40 | 43 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 8 | 8 | 19
  White | 46 | 42 | 47 | 135
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 39 | 44 | 45 | 128
  Germany | 15 | 9 | 12 | 36
Apnea-Hypopnea Index [Mean (Standard Deviation); unit: events/hour] — The Apnea-Hypopnea Index is the average number of apneas and hypopneas per hour of sleep during the routine clinical diagnostic polysomnography visit.
  events/hour | 36.87 (30) | 37.29 (31.1) | 41.08 (31.57) | 38.52 (30.6)

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index
Description: The Apnea-Hyopnea Index is the number of average number of apneas (complete pauses in breathing lasting at least 10 seconds) and hypopneas (decreases in airflow lasting at least 10 seconds) per hour of sleep. This data was compared from the polysomnography (sleep study) data after the first night of device use and at 180 days
Time Frame: Baseline and 180 Days
Population: During the course of the study 24 participants withdrew from the study.
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Auto Aflex | Auto CPAP | CPAP
Number analyzed (Participants) | 54 | 53 | 57
events/hour
  Baseline | 6.09 (7.20) | 3.54 (4.39) | 3.24 (3.46)
  180 Days: number analyzed (Participants) | 46 | 47 | 47
  180 Days | 1.26 (2.92) | 0.67 (0.93) | 1.04 (1.28)
Statistical Analysis 1: Comparison: Auto Aflex vs Auto CPAP vs CPAP; Test type: Superiority; p = 0.3, Kruskal-Wallis — PSG outcomes employed analysis of variance for approximately normally distributed outcomes (or outcomes that could be transformed to an approximately normal distribution), and the Kruskal-Wallis test for non-normal outcomes; Pairwise differences were determined using Tukey-Kramer test- ANOVA applied or by Mann-Whitney-Wilcoxon summed rank tests and Bonferroni adjustment

2. Secondary Outcome: Average Hours of Nightly Use.
Description: The average hours of nightly use is the average number of hours the participant used there device overnight at home during the study.
Time Frame: 180 days
Population: During the course of the study 24 participants withdrew from the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Auto Aflex | Auto CPAP | CPAP
Number analyzed (Participants) | 46 | 47 | 47
hours | 4.44 (1.98) | 4.63 (1.75) | 4.40 (2.02)

3. Secondary Outcome: Psychomotor Vigilance Task - Number of Lapses
Description: Psychomotor Vigilance Task-PVT is a 10-min attention/vigilance test. To measure trends of vigilance after 180 days of home use randomized sleep apnea trial. This measured how quickly participants reacted to visual stimulus and counted number of lapses.
  Lapses (errors of omission) are measured or usually defined as reaction Times ≥ 500 ms.
Time Frame: Baseline and 180 Days
Population: During the course of the study 24 participants withdrew from the study.
Measure: Mean (Standard Deviation); unit: number of lapses
Arm/Group | Auto Aflex | Auto CPAP | CPAP
Number analyzed (Participants) | 54 | 53 | 57
number of lapses
  Baseline | 2.15 (3.74) | 3.41 (7.75) | 2.15 (4.10)
  180 days: number analyzed (Participants) | 46 | 47 | 47
  180 days | 0.98 (2.14) | 0.96 (1.32) | 1.30 (3.32)

4. Secondary Outcome: Functional Outcomes of Sleep Questionnaire (FOSQ)
Description: FOSQ is a quality of life questionnaire for sleep disorders. It's a 30 question survey with 5 subgroups: general productivity (8 questions), social outcome (2 questions),activity level (9 questions), vigilance (7 questions) and intimate relationships & sexual activity (4 questions).
  Scores are provided on a 0 to 4 scale:
  0- I don't do this activity for other reasons or missing response
  1- Yes, extreme difficulty 4- no difficulty
  The average score was calculated based upon average sub-scores. The total score was,calculated using the mean of the subscale scores and multiplying the mean by the number of subscales. The range of scores for the total score is 5-20. The measures are designed to assess the impact of disorders of excessive sleepiness on activities of everyday living and the extent to which these abilities are improved by effective treatment. The lower the score the more difficulty a person has carrying out certain activities because they are too sleepy or tired.
Time Frame: Baseline and 180 Days
Population: During the course of the study 24 participants withdrew from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auto Aflex | Auto CPAP | CPAP
Number analyzed (Participants) | 54 | 53 | 57
score on a scale
  baseline | 15.17 (3.13) | 15.85 (2.94) | 14.57 (3.97)
  180 days: number analyzed (Participants) | 46 | 47 | 47
  180 days | 17.11 (2.22) | 17.78 (2.06) | 16.74 (3.26)

5. Secondary Outcome: Attitudes Toward Use
Description: Attitudes Toward Use Questionnaire (ATUQ) a self-efficacy scale based on psychological theories of behavior change and modified from one developed by Stepnowsky and Marler this outcome focused on confidence, expectations and importance.
  Confidence is a 5 question survey, it is measured on a scale of 1 to 5 1- disagree completely and 5 being agree completely. The scores range from 5 to 25 with 25 being extremely confident.
  Importance is a 11 question survey, it is measured on a scale of 1 to 5 1- disagree completely and 5 being agree completely. The importance ATU was combined with Exceptions survey, which is 4 questions. The expectations survey is measured on a scale of 1 to 5, with 1 being not at all effective and 5 extremely effective. The scores range from 15 to 75 with 75 being extremely important/ extremely effective.
Time Frame: Baseline and 180 Days
Population: During the course of the study 24 participants withdrew from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auto Aflex | Auto CPAP | CPAP
Number analyzed (Participants) | 54 | 53 | 57
units on a scale
  Confidence at baseline | 20.7 (3.6) | 21.8 (2.9) | 22.3 (2.6)
  Confidence at 180 days: number analyzed (Participants) | 46 | 47 | 47
  Confidence at 180 days | 20.7 (5.2) | 22.5 (3.3) | 21.9 (4.1)
  Expectations + Importance at baseline | 49.8 (7.4) | 48.4 (5.0) | 48.1 (6.9)
  Expectations + Importance at 180 days: number analyzed (Participants) | 46 | 47 | 47
  Expectations + Importance at 180 days | 47.2 (5.3) | 46.7 (5.8) | 46.9 (5.0)

6. Secondary Outcome: Subjective Assessment of Therapy Comfort.
Description: visual analog scales where used to assess the question "in the last month how do you rate the overall comfort of the mask"?
  0 = very uncomfortable to 100 = very comfortable
Time Frame: 30, 90, and 180 days
Population: During the course of the study 24 participants withdrew from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auto Aflex | Auto CPAP | CPAP
Number analyzed (Participants) | 54 | 53 | 57
units on a scale
  30 days: number analyzed (Participants) | 53 | 51 | 53
  30 days | 50.8 (21.5) | 57.9 (20.5) | 53.9 (18.9)
  90 days: number analyzed (Participants) | 51 | 46 | 51
  90 days | 53.8 (25.1) | 61.0 (15.0) | 59.2 (18.3)
  180 days: number analyzed (Participants) | 46 | 47 | 47
  180 days | 54.7 (21.7) | 60.1 (14.7) | 60.6 (17.9)

7. Secondary Outcome: Epworth Sleepiness Scale
Description: Epworth Sleepiness Scale is a test that measures sleepiness during daily life activities. This is an 8 question survey.
  Scores are provided on a 0 to 3 scale:
  0 = no chance of dozing
  1. = slight chance of dozing
  2. = moderate chance of dozing
  3. = high chance of dozing
  Scores range from 0 to 24. The higher the total number, the higher the overall sleepiness.
Time Frame: Baseline and 180 days
Population: During the course of the study 24 participants withdrew from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auto Aflex | Auto CPAP | CPAP
Number analyzed (Participants) | 54 | 53 | 57
units on a scale
  Baseline | 10.43 (5.25) | 10.49 (4.59) | 12.27 (5.94)
  180 Days: number analyzed (Participants) | 46 | 47 | 47
  180 Days | 6.93 (4.30) | 7.02 (4.66) | 7.87 (5.53)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Auto Aflex | Auto CPAP | CPAP
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/53 | 0/57
Other Adverse Events (participants affected / at risk) | 0/54 | 0/53 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No